CLINICAL TRIAL: NCT01637246
Title: A Study of Patients With Primary Open Angle Glaucoma or Ocular Hypertension Who Were Insufficiently Responsive to Monotherapy
Status: Completed | Type: Observational
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Other Study IDs: MAF/AGN/OPH/GLA/017; AGN-EPI-2009-02 (Other: Allergan)
Record Dates: First submitted 2012-07-09; First posted 2012-07-11 (Estimated); Results first posted 2012-09-21 (Estimated); Last update posted 2012-09-21 (Estimated); Status verified 2012-08

CONDITIONS: Glaucoma, Open-Angle; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- POAG or OHT: Patients with POAG or OHT previously treated with monotherapy and currently treated with any fixed combination therapy
  Interventions: Drug: Any Fixed Combination Therapy

INTERVENTIONS:
Drug: Any Fixed Combination Therapy — Patients with POAG or OHT previously treated with monotherapy and currently treated with any fixed combination therapy. This was a retrospective chart review study, so no treatment was administered in this study.

SUMMARY:
This is a retrospective chart review and will assess changes in IOP after treatment with any fixed combination in patients who previously received monotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of glaucoma or ocular hypertension
* Previously treated with monotherapy followed by fixed combination therapy for at least 12 weeks

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Primary Open Angle Glaucoma or Ocular Hypertension
Sampling Method: Non-Probability Sample
Enrollment: 4385 (Actual)
Dates: Start 2009-04; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Madrid, Spain

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | POAG or OHT
Started | 4385
Completed | 2246
Not Completed | 2139

BASELINE CHARACTERISTICS:
Arm/Group | POAG or OHT
Number analyzed (Participants) | 4385
Age Continuous [Mean (Standard Deviation); unit: Years]
  Data Available (N=2234) | 66.69 (11.43)
  Missing Data (N=2151) | NA (NA) — Age missing; not obtained
Sex/Gender, Customized [Number; unit: Participants]
  Female | 1177
  Male | 1111
  Missing Data | 2097

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Intraocular Pressure (IOP)
Description: IOP is a measurement of the fluid pressure inside the eye. A negative change from baseline indicates an improvement.
Time Frame: Baseline, 12 Weeks
Population: All patients who met the study entry criteria and have data for this outcome measure
Measure: Mean (Standard Deviation); unit: Millimeters of Mercury (mmHg)
Arm/Group | POAG or OHT
Number analyzed (Participants) | 2286
Millimeters of Mercury (mmHg)
  Baseline - Right Eye (N=2286) | 21.72 (3.62)
  Change from Baseline at 12 Wks-Rt Eye (N=2235) | -4.93 (3.24)
  Baseline - Left Eye (N=2248) | 21.59 (3.61)
  Change from Baseline at 12 Wks-Lft Eye (N=2192) | -4.88 (3.27)

2. Secondary Outcome: Patient Assessment of Tolerability Using a 4-Point Scale
Description: Patient assessment of tolerability using a 4-point scale (very good, good, moderate, and poor). The percentage of patients assessed as good and very good combined are reported.
Time Frame: 12 Weeks
Population: All patients who met the study entry criteria and have data for this outcome measure
Measure: Number; unit: Percentage of Patients
Arm/Group | POAG or OHT
Number analyzed (Participants) | 2244
Percentage of Patients | 79.2

3. Secondary Outcome: Physician Assessment of Tolerability Using a 4-Point Scale
Description: Physician assessment of tolerability using a 4-point scale (very good, good, moderate, and poor). The percentage of patients assessed as good and very good combined are reported.
Time Frame: 12 Weeks
Population: All patients who met the study entry criteria and have data for this outcome measure
Measure: Number; unit: Percentage of Patients
Arm/Group | POAG or OHT
Number analyzed (Participants) | 2307
Percentage of Patients | 87.6

4. Secondary Outcome: Percentage of Patients Who Maintained Better Compliance With Treatment
Description: Percentage of patients who maintained better compliance with treatment than prior therapy was assessed by the patient on a 3-point scale (better, equal, and worse compliance).
Time Frame: 12 Weeks
Population: All patients who met the study entry criteria and have data for this outcome measure
Measure: Number; unit: Percentage of Patients
Arm/Group | POAG or OHT
Number analyzed (Participants) | 2263
Percentage of Patients | 33.5

5. Secondary Outcome: Percentage of Patients Continuing on Therapy After 12 Weeks
Description: Percentage of patients continuing on therapy after 12 weeks was assessed as Yes or No.
Time Frame: 12 Weeks
Population: All patients who met the study entry criteria and have data for this outcome measure
Measure: Number; unit: Percentage of Patients
Arm/Group | POAG or OHT
Number analyzed (Participants) | 2265
Percentage of Patients | 92.9

ADVERSE EVENTS:
Arm/Group | POAG or OHT
Serious Adverse Events (participants affected / at risk) | 4/4385
Other Adverse Events (participants affected / at risk) | 0/4385
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | POAG or OHT (N=4385)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Keratitis (Eye disorders) | 2
Keratitis Herpetic (Eye disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No